CLINICAL TRIAL: NCT05880446
Title: PROstate CAncer Radiotherapy: Its Real Impact on Bowel Symptoms & Quality of Life Today, Measured by the EORTC QLQ C30 & Specific PRT20 Module.
Brief Title: PROstate CAncer Radiotherapy - Bowel Quality of Life (PROCAR-BQ)
Acronym: PROCAR-BQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Principal Investigator, Pauline De Bruyn, Principal Investigator, Jules Bordet Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IJB-PROCAR-BQ-2023; CE3650 (Other: Comité d'Ethique)
Record Dates: First submitted 2023-05-10; First posted 2023-05-30 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Prostate Cancer; Radiotherapy Side Effect; Bowel Dysfunction; Quality of Life
Keywords: Prostate Cancer; Radiotherapy Side Effect; Radiation Toxicity; Bowel Dysfunction; Pelvic Radiation Disease; Diarrhea; Radiation Proctitis; Radiation enteritis; Quality of Life; Malnutrition; Sarcopenia; Diet; Physical activity
MeSH Terms: conditions — Prostatic Neoplasms; Radiation Injuries; Intestinal Diseases; Diarrhea; Malnutrition; Sarcopenia; Motor Activity

STUDY DESIGN:
Intervention Model Description: Quality of life questionnaires and dietician advice before and at the end of treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bowel symptoms & QoL assessment (Other): This single arm study represent a group a patient with prostate cancer who are candidate for pelvic radiotherapy. Patient reported outcomes on bowel toxicity and overall quality of life will be systematically assessed right before and after RT. Various potential predictive factors will be analysed.
  Interventions: Other: Bowel symptoms & QoL assessment

INTERVENTIONS:
Other: Bowel symptoms & QoL assessment — QoL and bowel symptoms questionnaires will be held to patients, anthropomorphic measurement, handgrip test, physical activity level and usual diet quality of the patient will be assessed.

SUMMARY:
This is a prospective pilot study to evaluate the mean increase of bowel symptoms after pelvic radiotherapy (RT) in prostate cancer (PCa) patient using the validated & newly translated EORTC-QLQ PRT20 module.

DETAILED DESCRIPTION:
Questionnaires (QLQ-C30 and PRT20 modules) will be held to patients at the beginning and at the end of RT (4 weeks) to evaluate the mean increase of lower GI symptoms and decrease in overall QoL after pelvic RT.

For exploratory objectives, GLIM (Global Leadership Initiative on Malnutrition) criteria for malnutrition diagnosis, a 24h recall and DQI-I calculation will be assessed by the PI before the start of RT. CT sim & dosimetry will be analyse by the PI before treatment to evaluation the body composition and the max and mean dose received by the bowel, the sigmoid and the rectum. A Polar watches will be loaned to the patient by the PI at the CT sim appointment to record patient's daily movement for two weeks (usual waiting time between CT and treatment) and recovered on the first day of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men with PCa which are candidate for pelvic radiotherapy (RT) with or without previous surgery, with or without concomitant hormonotherapy (HT), Performance status (PS) 0-2 (all patient able to undergo RT treatment), of all age, elderly included.

Exclusion Criteria:

* Previous RT to the pelvis
* Diagnosed Inflammatory Bowel Disease (IBD), celiac disease
* Severe GI symptoms before the beginning of RT (Grade > 2 according to CTCAE grading system)
* Obvious cognitive impairment,
* Inability to understand French/English and no contact person able to accompany and translate.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-10-06 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
Mean Delta of EORTC Proctitis Module (PRT20) score | At study completion, an average of 4 months
  Mean Delta between the end and the beginning of RT (4 weeks) in PRT20 score (Min 18, Max 72, higher scores mean worse outcome)

SECONDARY OUTCOMES:
Mean Delta of EORTC Quality of Life Questionnaire (QLQ-C30) score | At study completion, an average of 4 months
  Mean Delta between the end and the beginning of RT (4 weeks) in C30 score (For symptoms: Min 28, Max 112, higher scores mean worse outcome; For general status: Min 2, Max 14, higher scores mean better outcome)

OTHER OUTCOMES:
Sarcopenia prevalence and its association with PRT20 and QLQ-C30 score Delta. | At study completion, an average of 4 months
  Descriptive analysis of sarcopenia prevalence and its association with PRT20 and QLQ-C30 score Delta.
  Men with L3 skeletal muscle index < 52.4 cm2/m2 will be classified as having sarcopenia. Skeletal muscle cross-sectional area (SMA) in cm2 at the third lumbar vertebra will be measured on the CT simulation (2 weeks before RT start) then normalized for stature to report the L3 skeletal muscle index (SMI) in cm2/m2. Hand-grip strength will be assessed as supportive measure the same day.
Malnutrition prevalence and its association with PRT20 and QLQ-C30 score Delta. | At study completion, an average of 4 months
  Descriptive analysis of GLIM (Global Leadership Initiative on Malnutrition) criteria for malnutrition diagnosis prevalence and its association with PRT20 and QLQ-C30 score Delta.
  One of the three positive phenotypic criteria will lead to positive diagnosis of malnutrition:
  * >5 % weight loss within past 6 months (asked to patient during visit or compared to previous reports),
  * BMI < 20-22 (weight and height will be combined to report BMI in kg/m^2),
  * Reduces muscle mass by L3 skeletal muscle index < 52.4 cm2/m2 (skeletal muscle cross-sectional area in cm2 at the third lumbar vertebra will be measured by CT then normalized for stature to report the L3 skeletal muscle index in cm2/m2)
Max Dose on Bowel Bag, Sigmoid & Rectum and its association with PRT20 and QLQ-C30 score Delta. | At study completion, an average of 4 months
  Descriptive analysis of Dmax in Gray (Gy) on Bowel Bag, Sigmoid & Rectum on RT plan dosimetry and its association with PRT20 and QLQ-C30 score Delta.
Mean Dose on Bowel Bag, Sigmoid & Rectum and its association with PRT20 and QLQ-C30 score Delta. | At study completion, an average of 4 months
  Descriptive analysis of Dmean in Gray (Gy) on Bowel Bag, Sigmoid & Rectum on RT plan dosimetry and its association with PRT20 and QLQ-C30 score Delta.
Low Diet Quality Index prevalence and its association with PRT20 and QLQ-C30 Delta | At study completion, an average of 4 months
  Descriptive analysis of Low Diet Quality Index (DQI-I) prevalence and its association with PRT20 and QLQ-C30 score Delta.
  DQI-I will be calculated from analysis of patient usual diet by the mean of a diet history and 24-h recall method before the start of RT and by it's conversion in nutritional values using composition tables. The continuous measure of the total DQI-I scores (Min 0, Max 100) of each patient will be categorized into quartiles (Very low, Low, Intermediate, High) and correlated to individual PRT20 and QLQ-C30 Delta in a descriptive manner.
Low Physical Activity Level prevalence and its association with PRT20 and QLQ-C30 Delta | At study completion, an average of 4 months
  Descriptive analysis of Low Physical Activity Level (PAL) prevalence and its association with PRT20 and QLQ-C30 score Delta.
  Physical Activity Level will be recorded by the mean of Polar® Watches which will be loaned to the patient by the PI at the CT sim appointment for two weeks (usual waiting time between CT and treatment) and recovered on the first day of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Jules Bordet, Anderlecht, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Delobel JB, Gnep K, Ospina JD, Beckendorf V, Chira C, Zhu J, Bossi A, Messai T, Acosta O, Castelli J, de Crevoisier R. Nomogram to predict rectal toxicity following prostate cancer radiotherapy. PLoS One. 2017 Jun 22;12(6):e0179845. doi: 10.1371/journal.pone.0179845. eCollection 2017. PMID 28640871
- [Background] Heemsbergen WD, Peeters ST, Koper PC, Hoogeman MS, Lebesque JV. Acute and late gastrointestinal toxicity after radiotherapy in prostate cancer patients: consequential late damage. Int J Radiat Oncol Biol Phys. 2006 Sep 1;66(1):3-10. doi: 10.1016/j.ijrobp.2006.03.055. Epub 2006 Jul 11. PMID 16814954
- [Background] Andreyev HJ, Benton BE, Lalji A, Norton C, Mohammed K, Gage H, Pennert K, Lindsay JO. Algorithm-based management of patients with gastrointestinal symptoms in patients after pelvic radiation treatment (ORBIT): a randomised controlled trial. Lancet. 2013 Dec 21;382(9910):2084-92. doi: 10.1016/S0140-6736(13)61648-7. Epub 2013 Sep 23. PMID 24067488
- [Background] Lawrie TA, Green JT, Beresford M, Wedlake L, Burden S, Davidson SE, Lal S, Henson CC, Andreyev HJN. Interventions to reduce acute and late adverse gastrointestinal effects of pelvic radiotherapy for primary pelvic cancers. Cochrane Database Syst Rev. 2018 Jan 23;1(1):CD012529. doi: 10.1002/14651858.CD012529.pub2. PMID 29360138
- [Background] Sini C, Noris Chiorda B, Gabriele P, Sanguineti G, Morlino S, Badenchini F, Cante D, Carillo V, Gaetano M, Giandini T, Landoni V, Maggio A, Perna L, Petrucci E, Sacco V, Valdagni R, Rancati T, Fiorino C, Cozzarini C. Patient-reported intestinal toxicity from whole pelvis intensity-modulated radiotherapy: First quantification of bowel dose-volume effects. Radiother Oncol. 2017 Aug;124(2):296-301. doi: 10.1016/j.radonc.2017.07.005. Epub 2017 Jul 21. PMID 28739383
- [Background] Halkett GKB, Wigley CA, Aoun SM, Portaluri M, Tramacere F, Livi L, Detti B, Arcangeli S, Lund JA, Kristensen A, McFadden N, Grun A, Bydder S, Sackerer I, Greimel E, Spry N; EORTC Quality of Life Group. International validation of the EORTC QLQ-PRT20 module for assessment of quality of life symptoms relating to radiation proctitis: a phase IV study. Radiat Oncol. 2018 Aug 29;13(1):162. doi: 10.1186/s13014-018-1107-x. PMID 30157890